CLINICAL TRIAL: NCT03585309
Title: The Impact of Electrocoagulation on Ovarian Reserve After Laparoscopic Excision of Ovarian Cysts: Randomization Clinical Trial
Brief Title: The Impact of Electrocoagulation on Ovarian Reserve After Laparoscopic Excision of Ovarian Cysts.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Zahra Hussein Mohammed Chewai, Resident of obstetrics and gynecology, Ain Shams University
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Ain shamsMH
Record Dates: First submitted 2018-05-07; First posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Ovarian Endometrioma; Ovary Cyst
MeSH Terms: conditions — Endometriosis; Ovarian Cysts

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparascopy comper with coagulation and without coagulation (Experimental)
  Interventions: Procedure: The impact of electrocoagulation on ovarian reserve after laparoscopic excision of ovarian cysts:

INTERVENTIONS:
Procedure: The impact of electrocoagulation on ovarian reserve after laparoscopic excision of ovarian cysts: — Randomization Randomization will be conducted using computer generated table. Group A (48 CASES) without coagulation
  Group A 6 89 92 35 1 15 21 16 60 49 53 91 34 5 94 64 88 58 7 33 8 75 29 56 10 23 37 19 32 71 55 84 36 77 50 2 46 70 82 9 51 54 72 18 25 31 14 63
  Group B (48 CASES) with coagulation Group B 79 38 93 43 52 44 62 47 68 76 86 95 81 83 42 80 94 30 78 61 12 17 66 13 41 59 22 73 39 65 4 90 28 26 3 87 40 85 69 48 27 24 74 57 11 20 67 45
  Allocation and concealment Nineteen six opaque envelopes will be numbered serially and in each envelope the corresponding letter which denotes the allocated group will be put according to randomization table then all envelopes will be closed and put in one box. When the first patient arrives the first envelope will be opened and the patient will be allocated according to the letter inside.

SUMMARY:
The aim of the study is to evaluate the effect of bipolar electrocoagulation on ovarian reserve.

DETAILED DESCRIPTION:
Laparoscopic ovarian cystectomy is currently considered the treatment of choice in women with benign ovarian cysts and has gained increasing acceptance among gynecologic sur¬geons . However, the safety of this technique in terms of ovarian damage to the operated gonad has recently been questioned. A great deal of evidence supports that the re¬moval of ovarian cysts is associated with injury to the ovarian reserve . Many of these studies involved patients who required assisted reproduction, and they found that the number both of follicles and retrieved oocytes obtained in the operated gonad during ovarian hyperstimulation was markedly reduced when compared with the contralateral intact ovary. However, most of these studies applied ovarian response to gonadotropin hyperstimulation to measure the ovarian reserve. It has been argued that these patients are not representative of all patients undergoing laparoscopic ovarian cystectomy in terms of ovarian damage because these data were acquired from aggressive gonadotropin stimulation which is thought to be different from a natural menstrual cycle .

On the other hand, because ovarian reserve cannot be mea¬sured directly, the evaluation of ovarian reserve is difficult to carry out. The induction of ovarian hyperstimulation in an un¬selected population of surgical patients for the purpose of evaluating ovarian reserve is obviously ethically untenable. The serum level of follicle-stimulating hormone (FSH) is a predictor of functional ovarian reserve , but its usefulness is limited considering that the vast majority of patients un¬dergo monolateral excision of a cyst and the contralateral in¬tact gonad may completely substitute for reduced function of the operated ovary . Given the well-established role of ul¬trasound scanning in the diagnosis and follow-up of ovarian cysts, reported that basal antral follicle number and mean ovarian diameter could be used as indicators of ovarian reserve. found that the value of ovarian stromal blood flow velocity was an initial marker of ovarian reserve before the change of FSH level and ovarian volume.

With the combined use of serum hormonal evaluation and ultrasound examination, the investigators prospectively investigated the ovarian reserve of patients after the excision of benign ovarian cysts. The damage to ovarian reserve was evaluated during through a 12-month follow-up period after the application of bipolar, ultrasonic scalpel electrocoagulation or suture for ovarian cystectomy .

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-35 years.
2. Uni-bilateral ovarian cyst(s) size without clinical and sonographic suspicion of ovarian cancer.
3. Regular menstrual cycles defined as a cycle length between 25 and 35 days in the 6 months before surgery.
4. Agreement to be enrolled in the study.
5. Endometriosi.
6. Renal disesase.
7. Liver disease.

Exclusion Criteria:

* 1- Prior ovarian surgery 2- Surgical necessity to perform adnexectomy 3- Known endocrine disease 4- Postoperative pathologic diagnosis that was not benign ovarian cyst 5- Oral contraceptive use before surgery last two months. 6-Addison disease. 7.Thyroid disease.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 96 (Estimated)
Dates: Start 2018-07-15 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants (Females) with ovarian cyst or dermid cyst or endometrial | 3 months after surgery
  Laparascopy without coagulation excision of ovarian cysts and effect of ovarian reserve RESULIT The result of the study is to evaluate the effect of bipolar electrocoagulation on ovarian reserve.

SECONDARY OUTCOMES:
Number of participants (Females) with ovarian cyst or dermid cyst or endometrial | 3 months after surgery
  Laparascopy with coagulation excision of ovarian cysts and effect of ovarian reserve RESULT The result of the study is to evaluate the effect of bipolar electrocoagulation on ovarian reserve.

CONTACTS AND LOCATIONS:
Overall Officials: kareem labib, MD, Principal Investigator — Ain shams University Maternity Hospital
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

REFERENCES:
- [Background] Asgari Z, Rouholamin S, Hosseini R, Sepidarkish M, Hafizi L, Javaheri A. Comparing ovarian reserve after laparoscopic excision of endometriotic cysts and hemostasis achieved either by bipolar coagulation or suturing: a randomized clinical trial. Arch Gynecol Obstet. 2016 May;293(5):1015-22. doi: 10.1007/s00404-015-3918-4. Epub 2015 Oct 22. PMID 26493551